CLINICAL TRIAL: NCT02130817
Title: Belatacept for the Management of Moderately Sensitized Patients at Risk for Delayed Graft Function (DGF)
Brief Title: Belatacept in Kidney Transplantation of Moderately Sensitized Patients
Acronym: BelatPilot
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Organ transplant criteria made recruitment difficult. Closed with IRB 10/09/2015.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Should be 2013-0672; IM103-327 (Other: Study Team)
Record Dates: First submitted 2014-04-30; First posted 2014-05-05 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: End Stage Renal Disease; Antibody Mediated Rejection
Keywords: Renal Transplant; Kidney Transplant; Mean flourescent Intensity; Delayed Graft Function; Antagonist of Thymocyte Cell Activation
MeSH Terms: conditions — Kidney Failure, Chronic; Delayed Graft Function | interventions — Abatacept; Plasmapheresis; thymoglobulin; Antilymphocyte Serum; Mycophenolic Acid; Steroids; Dexamethasone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Belatacept (Experimental): Belatacept (nujolix):
  Tacrolimus withdrawal
  Standard of care(SOC) treatment:
  Plasmapheresis/Intravenous Immunoglobulin G (IVIG) therapy
  Thymoglobulin will be administered to a total cumulative dose of 4.5-6 mg/kg starting in the operating room.
  Maintenance immunosuppression:
  Myfortic: Patients will receive 720mg bid of Myfortic throughout the study, starting day 1 after surgery.
  Steroids: Patients will receive Dexamethasone IV on the day of surgery (Day 0) with tapered doses through Day 4 followed by prednisone tapered to 10mg/d by day 30.
  Interventions: Drug: Belatacept; Drug: Tacrolimus withdrawal; Procedure: Plasmapheresis/Intravenous Immunoglobulin G; Drug: Thymoglobulin (ATG); Drug: Myfortic; Drug: Steroids

INTERVENTIONS:
Drug: Belatacept — Belatacept will be added to the standard of care regimen and will be given at days 0,5, weeks 2, 4, 8 and 12 (10 mg/kg) and every 4 weeks (5 mg/kg) for one year.
  Other Names: Nujolix
Drug: Tacrolimus withdrawal — Tacrolimus dosing will begin on Days 1 through 5 post transplant at up to 2 mg BID to achieve target trough levels of 9-11 ng/ml. The dose will be tapered through the end of week 2 to achieve a trough level of 4 ng/ml which will be maintained for six weeks. Tacrolimus will be withdrawn at the end of eight weeks post transplant.
Procedure: Plasmapheresis/Intravenous Immunoglobulin G — Enrolled patients will start with standard of practice treatment including plasmapheresis and IVIG therapy twice after transplant, on days 2 and 4 and potentially once before transplant. Plasmapheresis and albumin exchange for one volume of blood will be performed in the infusion center at the University of Wisconsin Hospital and Clinics (UWHC). Each pheresis session will be completed by IVIG infusion. While plasmapheresis will help with the removal of circulating Donor Specific Antibodies (DSA), IVIG therapy will provide immunomodulatory characteristics that include sterilizing immunity from infections, inhibiting and scavenging activated complement fragments, modifying cell-mediated immune responses, inducing regulatory T cells and importantly, inhibiting deleterious antibody production.
Drug: Thymoglobulin (ATG) — Thymoglobulin (ATG) Induction. Thymoglobulin will be administered to a total cumulative dose of 4.5-6 mg/kg via a peripheral or central vein, starting in the operating room.
  Other Names: Anti-thymocyte globulin
Drug: Myfortic — Patients will receive 720mg bid of Myfortic throughout the study, starting day 1 after surgery.
Drug: Steroids — Patients will receive Dexamethasone IV on the day of surgery (Day 0) with tapered doses through Day 4 followed by prednisone tapered to 10mg/d by day 30.,
  Other Names: Dexamethasone, Prednisone

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an immunosuppressive medication, Belatacept, as a replacement for a calcineurin inhibitor, in combination with a standard of care regimen of immunosuppressive medications and plasma exchange (plasmapheresis and immunoglobulin treatment) for kidney transplant patients who are moderately sensitized against their deceased donor and at-risk for delayed graft function. The hypothesis is that moderately sensitized patients who receive Belatacept treatment with the standard of care regimen will lead to lower acute rejection rates than historical controls based on assessment of standard of care biopsies and standard Banff criteria.

DETAILED DESCRIPTION:
This exploratory single-center, open-label safety and efficacy study will enroll 20 adult kidney transplants candidates, moderately sensitized against their deceased donor and at-risk for delayed graft function (DGF), to receive Belatacept (days 0,5, weeks 2,4,8 and 12 (10 mg/kg), and every 4 weeks thereafter (5 mg/kg)), plasma exchange (once before and twice after transplant) and Intravenous Immunoglobulin (IVIG) (100 mg/kg after each plasma exchange), along with Thymoglobulin (ATG) induction and Dexamethasone tapered dosing starting on the day of transplant at 100mg IV, tapered through Day 4, followed by prednisone at 30 mg on Day 5 with tapered dosing to prednisone 10 mg/d by one month, with a total observation period of 1 year. Patients will be tapered off tacrolimus by week 8 and will remain on mycophenolic acid and prednisone for the total length of the study. Subjects will be followed until 1 year post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18-70 years of age
* Patient who is receiving an expanded criteria donor (ECD) or deceased cardiac donor (DCD) kidney
* Have immunodominant donor specific antibodies (DSA) 1,000 - 4,000 mean fluorescent intensity (MFI) by single bead Luminex bioassay
* Subjects must be capable of understanding the investigational nature and risks of the study and must sign a statement of informed consent
* Female patients of child bearing potential must have a negative urine or serum pregnancy test within the past 48 hours prior to study inclusion and be willing to use contraceptives for the duration of the study and for 8 weeks after the last dose of study drug Women of Child-Bearing Potential (WOCBP) includes
* Women who have experienced menarche and who have not undergone successful surgical sterilization or who are not post-menopausal
* Women using oral contraceptives, other hormonal contraceptives, or mechanical products such as intrauterine devices or barrier methods
* Women who are practicing abstinence
* Women who have a partner who is sterile (eg, due to vasectomy).
* Women must not be breast-feeding
* Male subjects must agree to use an acceptable method for contraception for the duration of the study
* Patient must have known positive Epstein-Barr virus (EBV) serostatus

Exclusion Criteria:

* Patient has previously received an organ transplant other than a kidney.
* Patient is receiving an human leukocyte antigen (HLA) identical living donor transplant
* Patient who is a recipient of a multiple organ transplant
* Patient with a positive T or B cell crossmatch
* Patient with a donor specific antibody (DSA) as deemed by the local PI to be associated with significant risk of rejection
* Patient has received an ABO incompatible donor kidney
* Recipients will be receiving a dual or en bloc kidney transplant
* Donor anticipated cold ischemia is > 30hours
* Recipient or donor is known to be seropositive for hepatitis C virus (HCV) or B virus (HBV) except for hepatitis B surface antibody positive. HCV seropositive patients with a negative HCV viral load testing may be included.
* Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV)
* Seronegative or unknown EBV serostatus
* Patient has uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives
* Patients with tuberculosis who have not been treated for latent infection.
* Patients at high risk for polyoma virus-associated nephropathy, which is mostly due to BK virus infection
* Patients at high risk for polyoma virus-associated nephropathy, which is mostly due to BK virus infection
* Patients with thrombocytopenia (PLT <75,000/mm3), and/or leucopoenia (WBC < 2,000/mm3), or anemia (hemoglobin < 6 g/dL) prior to study inclusion.
* Patient is taking or has been taking an investigational drug in the 30 days prior to transplant
* Patient who has undergone desensitization therapy within 6 months prior to transplant
* Patient has a known hypersensitivity to belatacept, tacrolimus, mycophenolate mofetil, alemtuzumab, rabbit anti-thymocyte globulin, or glucocorticoids
* Patient is receiving chronic steroid therapy at the time of transplant
* Patients with a history of cancer (other than non-melanoma skin cell cancers cured by local resection) within the last 5 years
* Patients with > Grade 2 peripheral neuropathy within 14 days before enrollment
* Myocardial infarction within 6 months prior to enrollment or New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiography evidence of acute ischemia or active conduction system abnormalities.
* Female subject is pregnant or breast-feeding
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study. Subjects who are compulsorily detained for treatment of either a psychiatric or physical illness
* Prisoners or subjects who are involuntarily incarcerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2015-10-09 (Actual); Study Completion 2015-10-09 (Actual)

PRIMARY OUTCOMES:
Acute rejection | one year
  Acute rejection rates are based on assessment of standard of care biopsy (protocol and indication) and standard Banff criteria.

SECONDARY OUTCOMES:
Patient and Graft Survival | One year
  The number of subjects alive and with functioning grafts at one year.
Incidence of infections | One year
  Number of subjects in the study who have developed infections, including cytomegalovirus (CMV) and BK Virus, in the first year post-transplant
Incidence of de novo donor specific antibody (DSA) | One year
  Number of subjects who have developed donor specific antibodies at one year post transplant.
Incidence of new onset diabetes | One year
  Number of subjects in the study who have developed new onset diabetes since receiving the transplant
Increase in estimated Glomerular Filtration Rate (eGFR) | One year
  Number of subjects in the study whose eGFR has decreased to < 45 milliliters/ minute
Incidence of malignancies | One year
  Number of subjects in the study who have developed malignancies including post-transplant lymphoproliferative (PTLD) disorder

CONTACTS AND LOCATIONS:
Overall Officials: Arjang Djamali, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wiscsonsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Trivedi HL, Terasaki PI, Feroz A, Everly MJ, Vanikar AV, Shankar V, Trivedi VB, Kaneku H, Idica AK, Modi PR, Khemchandani SI, Dave SD. Abrogation of anti-HLA antibodies via proteasome inhibition. Transplantation. 2009 May 27;87(10):1555-61. doi: 10.1097/TP.0b013e3181a4b91b. PMID 19461494
- [Background] Jordan SC, Pescovitz MD. Presensitization: the problem and its management. Clin J Am Soc Nephrol. 2006 May;1(3):421-32. doi: 10.2215/CJN.01651105. Epub 2006 Apr 12. PMID 17699241
- [Background] Stegall MD, Gloor J, Winters JL, Moore SB, Degoey S. A comparison of plasmapheresis versus high-dose IVIG desensitization in renal allograft recipients with high levels of donor specific alloantibody. Am J Transplant. 2006 Feb;6(2):346-51. doi: 10.1111/j.1600-6143.2005.01178.x. PMID 16426319
- [Background] Vo AA, Lukovsky M, Toyoda M, Wang J, Reinsmoen NL, Lai CH, Peng A, Villicana R, Jordan SC. Rituximab and intravenous immune globulin for desensitization during renal transplantation. N Engl J Med. 2008 Jul 17;359(3):242-51. doi: 10.1056/NEJMoa0707894. PMID 18635429
- [Background] Montgomery RA, Zachary AA. Transplanting patients with a positive donor-specific crossmatch: a single center's perspective. Pediatr Transplant. 2004 Dec;8(6):535-42. doi: 10.1111/j.1399-3046.2004.00214.x. PMID 15598320
- [Background] Magee CC, Felgueiras J, Tinckam K, Malek S, Mah H, Tullius S. Renal transplantation in patients with positive lymphocytotoxicity crossmatches: one center's experience. Transplantation. 2008 Jul 15;86(1):96-103. doi: 10.1097/TP.0b013e318176ae2c. PMID 18622284
- [Background] Thielke JJ, West-Thielke PM, Herren HL, Bareato U, Ommert T, Vidanovic V, Campbell-Lee SA, Tzvetanov IG, Sankary HN, Kaplan B, Benedetti E, Oberholzer J. Living donor kidney transplantation across positive crossmatch: the University of Illinois at Chicago experience. Transplantation. 2009 Jan 27;87(2):268-73. doi: 10.1097/TP.0b013e3181919a16. PMID 19155983
- [Background] Jordan SC, Toyoda M, Vo AA. Intravenous immunoglobulin a natural regulator of immunity and inflammation. Transplantation. 2009 Jul 15;88(1):1-6. doi: 10.1097/TP.0b013e3181a9e89a. PMID 19584672
- [Background] Investigator Brochure. Belatacept (BMS-2224818), Version 13. Bristol-Myers Squibb Research and Development Department. 15 December 2010.
- [Background] U.S. Prescribing information for Nulojix® (belatacept), Revised 06/2011. Bristol-Myers Squibb.